CLINICAL TRIAL: NCT00350285
Title: Reaching and Motivating Change in Teen Marijuana Smokers
Brief Title: The Teen Marijuana Check-Up
Acronym: TMCU3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Roger A. Roffman /Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-8666-G-05; R01DA014296 (NIH)
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Cannabis Abuse; Cannabis Dependence
Keywords: cannabis; marijuana
MeSH Terms: conditions — Marijuana Abuse | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Motivational enhancement therapy
  Interventions: Behavioral: Motivational enhancement therapy
- 2 (Active Comparator): Marijuana education
  Interventions: Behavioral: Marijuana education
- 3 (No Intervention): Delayed treatment control condition

INTERVENTIONS:
Behavioral: Motivational enhancement therapy — Personal feedback with counselor using motivational interviewing strategies.
  Arms: 1
Behavioral: Marijuana education — Information about health and behavioral effects of marijuana use.
  Arms: 2

SUMMARY:
This behavioral research is an efficacy trial evaluating an intervention called "The Teen Marijuana Check-Up" with non-treatment seeking adolescent marijuana users.

DETAILED DESCRIPTION:
Three hundred adolescents who smoke marijuana (ages 14-19), recruited in four Seattle-area high schools, will be enrolled in the trial. Participants will be recruited either through in-class presentations focusing on marijuana or via referrals from school staff. They will first be assessed regarding use of marijuana, alcohol, and other drugs, as well as pertinent attitudes and goals. Participants will then be randomly assigned to one of three conditions.

* The experimental intervention is a two-session motivational enhancement treatment. A personalized feedback report, containing information from the participant's assessment as well as normative comparison data, is reviewed, with the Health Educator employing motivational interviewing strategies intended to enhance motivation for reduction or cessation of marijuana use. Specific goals for change and behavior change strategies are discussed with participants who wish support to change their marijuana use.
* The comparison condition involves two educational sessions focusing on the health and behavioral effects of marijuana.
* The third condition (delayed treatment control) involves a minimal baseline assessment followed three months later by a reassessment interview. Those assigned to this condition will then be given their choice of either active treatment.

Following completion of their two intervention sessions, participants in the two active treatments will be offered an additional four sessions of cognitive-behavioral skills training in which the focus is strategies in quitting marijuana. All participants will be reassessed at 3 and 12 months following their initial assessment interviews.

ELIGIBILITY:
Inclusion Criteria: Individuals who contact the project will be screened according to the following inclusion criteria:

* age (14-19 years old),
* grade level (freshmen through seniors) and
* marijuana use (smoked 9 or more days in past 30).

Exclusion Criteria: Individuals will be excluded if:

* they are not fluent in English,
* they have a thought disorder that precludes full participation,
* they refuse to accept randomization to condition.

In addition to the inclusion and exclusion criteria, participants who appear to be in psychological or physical distress will be assessed further and referred to other services as appropriate. The need for other services will not necessarily preempt participation in the TMCU unless the individual is incapable or unwilling to complete the protocol. As was the case in our Stage 1b trial, all ineligible applicants will be offered a single feedback session, and the Strategies That Work booklet will be offered to those who indicate any interest in reducing or quitting marijuana use.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 310 (Actual)
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Self-report of marijuana use | 3 months and 12 months

SECONDARY OUTCOMES:
Accepting abstinence-focused counseling | 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roger A Roffman, DSW, Principal Investigator — University of Washington School of Social Work